CLINICAL TRIAL: NCT04823949
Title: Remote Monitoring Compared With In-Office Surveillance of Blood Pressures in Patients With Pregnancy-Related Hypertension: A Randomized Controlled Trial
Brief Title: Pregnancy-Related Hypertension: Adherence to a New Type of Monitoring
Acronym: PHANTOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Medical University of South Carolina (Other); South Carolina Telehealth Alliance (Other); Babyscripts (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00090951
Record Dates: First submitted 2020-12-03; First posted 2021-04-01 (Actual); Results first posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-04

CONDITIONS: Gestational Hypertension; Preeclampsia; Chronic Hypertension With Pre-Eclampsia Complicating Childbirth; HELLP Syndrome
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Pre-Eclampsia; HELLP Syndrome | interventions — Blood Pressure Monitoring, Ambulatory

STUDY DESIGN:
Intervention Model Description: Control arm: will be scheduled an in-office blood pressure check 7-10 days postpartum Intervention arm: will receive a blood pressure cuff and app with which to monitor their blood pressures at home for 16 days postpartum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard care (No Intervention): Patient will be scheduled for a blood pressure check in the office 7-10 days postpartum
- Intervention (Experimental): Patient will receive a Babyscripts blood pressure cuff(brand: A&D Medical) and Babyscripts MyJourney phone app with which to monitor their blood pressures twice daily for 16 days after discharge
  Interventions: Device: Home blood pressure monitoring

INTERVENTIONS:
Device: Home blood pressure monitoring — See arm description
  Arms: Intervention

SUMMARY:
A large segment of our patient population is diagnosed with hypertensive disorders of pregnancy, including gestational hypertension and pre-eclampsia. New guidelines from the American College of Obstetricians and Gynecologists recommend postpartum monitoring of blood pressures via blood pressure checks on day 3 postpartum and between days 7-10 postpartum. Our purpose is to compare the effectiveness of using a Bluetooth-enabled home blood pressure monitoring platform to the standard postpartum office-based blood pressure monitoring in performing the recommended postpartum follow-up for patients with hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
While inpatient during the postpartum period, patients will be identified who were diagnosed with hypertensive disorders of pregnancy antepartum, intrapartum, or postpartum. These patients will be recruited prior to discharge home. This will be a randomized control trial, non-blinded. The study group will receive a mobile app for postpartum education and an integrated Wi-Fi connected blood pressure cuff for at-home monitoring for 16 days postpartum. The home BP monitoring will occur twice a day and study team will check the BPs twice a day and intervene by phone or text if necessary. The control group will be scheduled for blood pressure checks at the clinic between days 7-10. These groups will be compared with regard to adherence to guidelines from the American College of Obstetricians and Gynecologists for blood pressure monitoring, antihypertensive initiation after discharge, unscheduled visits, readmission, and attendance of postpartum visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have delivered an infant either at Greenville Memorial Hospital or MUSC and be willing and able to follow-up with her respective institution.
* Patient must have been diagnosed with a hypertensive disorder of pregnancy in the antepartum, intrapartum, or postpartum period.

Exclusion Criteria:

* <18 years of age
* BMI >50 (due to limitations in blood pressure cuff size through BabyScripts)
* non English-speaking
* not able to receive phone calls and unlimited texts on cell phone
* not able to download and use Babyscripts phone application

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renata Sawyer, MD, Principal Investigator — Prisma Health-Upstate; David Soper, MD, Principal Investigator — Medical University of South Carolina
Locations (2):
- United States (2):
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arkerson BJ, Finneran MM, Harris SR, Schnorr J, McElwee ER, Demosthenes L, Sawyer R. Remote Monitoring Compared With In-Office Surveillance of Blood Pressure in Patients With Pregnancy-Related Hypertension: A Randomized Controlled Trial. Obstet Gynecol. 2023 Oct 1;142(4):855-861. doi: 10.1097/AOG.0000000000005327. Epub 2023 Sep 7. PMID 37734091

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was conducted at Prisma Health (Greenville, SC, USA) and the Medical University of South Carolina (Charleston, SC, USA) between April 2021 and September 2021.
  The recruitment took place inpatient at the obstetric units of both hospitals.
Groups:
- Standard Care: Patient will be scheduled for a blood pressure check in the office within 10 days of the postpartum discharge
- Intervention: Patient will receive a Babyscripts blood pressure cuff (brand: A&D Medical) and Babyscripts MyJourney phone app with which to monitor their blood pressures twice daily for 16 days after discharge
  Home blood pressure monitoring: See arm description
Period: Overall Study
Arm/Group | Standard Care | Intervention
Started | 101 | 101
Completed | 101 | 96
Not Completed | 0 | 5
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | Intervention | Total
Number analyzed (Participants) | 101 | 96 | 197
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.6 [23.2 to 33.6] | 28.9 [23.7 to 32.2] | 29.1 [23.3 to 32.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 96 | 197
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 34 | 28 | 62
  White | 59 | 56 | 115
  Asian | 3 | 0 | 3
  Hispanic | 4 | 11 | 15
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 101 | 96 | 197
Insurance [Count of Participants; unit: Participants]
  Private | 39 | 36 | 75
  Medicaid | 58 | 59 | 117
  None | 4 | 1 | 5
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 34.0 [26.6 to 39.3] | 32.9 [26.2 to 39.6] | 33.3 [26.4 to 39.5]
Tobacco use [Count of Participants; unit: Participants]
  None | 59 | 68 | 127
  Former | 28 | 16 | 44
  Current | 13 | 12 | 25
  Unknown | 1 | 0 | 1
Chronic Hypertension [Count of Participants; unit: Participants] | 26 | 17 | 43
Diabetes [Count of Participants; unit: Participants]
  Gestational diabetes | 10 | 20 | 30
  Type 2 Diabetes | 2 | 5 | 7
  Type 1 Diabetes | 2 | 1 | 3
Renal Disease [Count of Participants; unit: Participants] | 11 | 11 | 22
Timing of Diagnosis [Count of Participants; unit: Participants]
  Antepartum | 70 | 57 | 127
  Intrapartum | 25 | 29 | 54
  Postpartum | 6 | 10 | 16
Gestational Age at Delivery [Median (Inter-Quartile Range); unit: Weeks] | 37.3 [34.1 to 38.7] | 37.5 [34.5 to 39.1] | 37.3 [34.4 to 39]
Hypertensive Disease Severity [Count of Participants; unit: Participants]
  Gestational hypertension | 37 | 42 | 79
  Preeclampsia without severe features | 15 | 7 | 22
  Preeclampsia with severe features | 48 | 43 | 91
  HELLP syndrome | 0 | 2 | 2
  Eclampsia | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Adherence to the American College of Obstetricians and Gynecologists Guideline of Postpartum Blood Pressure Check Within 10 Days Postpartum
Description: How many participants had a blood pressure check within 10 days postpartum as recommended by the American College of Obstetricians and Gynecologists
Time Frame: 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 101 | 96
Participants | 59 | 89
Statistical Analysis 1: Comparison: Standard Care vs Intervention; Test type: Other; p < 0.001, Chi-squared; Risk Ratio (RR) = 1.59, 95% CI 2-sided [1.33 to 1.88]

2. Secondary Outcome: Initiation of Antihypertensive After Discharge
Description: How many participants required initiation of antihypertensive after discharge
Time Frame: 16 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 101 | 96
Participants | 7 | 9
Statistical Analysis 1: Comparison: Standard Care vs Intervention; Test type: Other; p = .530, Fisher Exact; Risk Ratio (RR) = 1.35, 95% CI 2-sided [0.52 to 3.49]

3. Secondary Outcome: Unscheduled Visits
Description: Number of participants with unscheduled visits
Time Frame: 16 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 101 | 96
Participants | 5 | 12
Statistical Analysis 1: Comparison: Standard Care vs Intervention; Test type: Other; p = .059, Fisher Exact; Risk Ratio (RR) = 2.53, 95% CI 2-sided [0.92 to 6.90]

4. Secondary Outcome: Readmission
Description: Number of participants readmitted postpartum
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 101 | 96
Participants | 5 | 4
Statistical Analysis 1: Comparison: Standard Care vs Intervention; Test type: Other; p = .792, Fisher Exact; Risk Ratio (RR) = 0.84, 95% CI 2-sided [0.23 to 3.04]

5. Secondary Outcome: Attended Postpartum Visit
Description: Number of participants who attended their postpartum visit
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Care | Intervention
Number analyzed (Participants) | 101 | 96
Participants | 71 | 75
Statistical Analysis 1: Comparison: Standard Care vs Intervention; Test type: Other; p = .210, Chi-squared; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.94 to 1.31]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Standard Care | Intervention
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/101
Other Adverse Events (participants affected / at risk) | 0/101 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT04823949/Prot_002.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT04823949/SAP_003.pdf
  • Informed Consent Form (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT04823949/ICF_004.pdf